CLINICAL TRIAL: NCT02549989
Title: Single-Arm, Open-Label, Phase II Study of LY3023414 for the Treatment of Recurrent or Persistent Endometrial Cancer
Brief Title: Study of LY3023414 for the Treatment of Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-079
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-03

CONDITIONS: Endometrial Cancer; Recurrent Endometrial Cancer
Keywords: LY3023414; 15-079; Persistent Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — LY3023414

ARMS (1):
- LY3023414 (Experimental): This is an MSKCC investigator-initiated, single-center, non-randomized, open-label, phase II study to evaluate the activity of LY3023414 dosed at the RP2D of 200 mg orally twice daily in patients with recurrent or persistent endometrial cancer.
  Interventions: Drug: LY3023414

INTERVENTIONS:
Drug: LY3023414 — Enrolled patients will take LY3023414 200 mg orally twice a day. Each cycle will be 21 days in duration. Patients will receive study treatment until disease progression, intolerable toxicity, elective withdrawal from the study, study completion, or study termination

SUMMARY:
The purpose of this study is to determine the effectiveness of LY3023414 in treating the participants type of cancer and to determine the types and severity of side effects caused by treatment with LY3023414.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, transitional cell carcinoma, and carcinosarcoma.
* Age ≥ 18 years
* Patients must have had at least one but no more than four prior chemotherapeutic regimens for management of endometrial carcinoma (including neo-adjuvant and/or adjuvant chemotherapy). Initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen.
* Patients tumors must have known PI3K pathway activation defined as EITHER of the following on a CLIA-approved molecular diagnostics test:
* Genomic alteration resulting in loss of PTEN function including a) whole or partial gene deletion, frame shift mutations, or non-sense mutations. Missense mutations in PTEN will not be considered qualifying.
* A previously characterized activating mutation in any component of the pathway including: PIK3CA, AKT1, PIK3R1, PIK3R2, mTOR
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Resolution of adverse effects of recent surgery, radiotherapy, or chemotherapy to Grade ≤1 prior to first study treatment (with the exception of alopecia or neuropathy).
* Patients must have measurable disease. Measurable disease is defined by RECIST (version 1.1). Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or ≥ 20 mm when measured by chest x-ray. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI.
* No active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection).
* Any other prior therapy directed at the malignant tumor, including immunologic agents and radiotherapy, must be discontinued at least 2 weeks prior to first study treatment.
* Adequate hematologic defined by the following laboratory results obtained within 14 days prior to first study treatment:
* Absolute neutrophil count (ANC) ≥1500/10^9dL
* Platelet count ≥ 100,000/10^9dL
* Hemoglobin ≥ 9.0 g/dL
* Adequate hepatic function defined by the following laboratory results obtained within 14 days prior to first study treatment:
* Total bilirubin≤1.5x the upper limit of normal (ULN)
* AST and ALT ≤ 3.0x ULN (unless the patient has Gilbert's Syndrome, in which case AST and ALT ≤ 5.0x ULN is permitted
* Albumin ≥ 3.5 g/dL
* Adequate renal function defined by the following laboratory results obtained within 14 days prior to first study treatment:
* Serum creatinine≤1.5x ULN OR creatinine clearance ≥50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation
* For all patients (regardless of known diabetes) the following is required at screening: Fasting blood glucose ≤ 135 mg/dL (7.49 mmol/L) and HbA1c ≤7.0%
* For patients of childbearing potential, agreement to use two effective forms of contraception (e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) and to continue its use for the duration of the study and for 30 days after the last LY3023414 dose.
* Patients must have been enrolled, or agree to consent to the companion genomic profiling study MSKCC IRB# 12-245.
* Willingness to sign written informed consent to this study.

Exclusion Criteria:

* Patients with known concurrent activating RAS/RAF mutation or loss of function mutation or deletion in NF1 of NF2 resulting in MAP kinase pathway activation. Patients are not required to be evaluated for these alterations if not already performed.
* Patients with diabetes requiring insulin or requiring more than one non-insulin hypoglycemia agents.
* Patients previously treated with an mTOR, AKT, or PI3K inhibitor (including but not limited to GDC-0941, GDC-0980, BEZ235, BKM120, LY294002, PIK-75, TGX-221, XL147, XL765, SF1126, PX-866, D-87503, D-106669, GSK615, CAL101, everolimus, temsirolimus, and ridaforolimus). For agents not listed, the Study PI or Co-PI will make a determination.
* History of myocardial infarction or unstable angina within 6 months prior to first study treatment.
* New York Heart Association Class II or greater congestive heart failure.
* Patients with a QTcF interval of >450 msec on screening electrocardiogram (ECG) Note: If >450 msec on the first ECG, 2 additional ECGs can be ordered same day and then the average may be used to determine eligibility.
* History of malabsorption syndrome or other condition that would interfere with enteral absorption.
* Inability or unwillingness to swallow pills
* Clinically significant history of liver disease, including cirrhosis and current alcohol abuse.
* Active hepatitis B or hepatitis C infection. Patients with previously resolved hepatitis B infection are eligible. Presence of positive test results for hepatitis B infection who have resolved the infection (defined by being positive for HB surface antibody (anti-HBs) and polymerase chain reaction (PCR) assay is negative for HBV DNA) are eligible. Patients positive for HCV antibody are eligible only if testing for HCV RNA is negative.
* Known HIV infection.
* Need for current chronic corticosteroid therapy (≥ 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids)
* Pregnancy, lactation, or breastfeeding
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1 or anticipation of the need for major surgery during the course of study treatment.
* Known untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided that they meet all of the following criteria:
* Presence of measurable disease outside the CNS
* No radiographic evidence of worsening upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
* No history of intracranial hemorrhage or spinal cord hemorrhage
* No ongoing requirement for dexamethasone as therapy for CNS disease (anticonvulsants at a stable dose are allowed)
* Absence of leptomeningeal disease
* Inability to comply with study and follow-up procedures.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Makker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY3023414
Started | 28
Completed | 1
Not Completed | 27
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Lack of Efficacy | 19
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | LY3023414
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 65 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: defined as the percentage of patients with complete response (CR) + partial response (PR) + stable disease (SD) ≥12 weeks from the start of treatment.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 12 weeks from baseline up to a year
Measure: Count of Participants; unit: Participants
Arm/Group | LY3023414
Number analyzed (Participants) | 25
Participants
  Participants with Clinical Benefit Rate (CR+PR+SD) | 7
  Participants without CBR | 18

2. Primary Outcome: Overall Response Rate
Description: determined by RECIST 1.1.
Time Frame: 1 year
Measure: Mean (90% Confidence Interval); unit: percentage of participants
Arm/Group | LY3023414
Number analyzed (Participants) | 28
percentage of participants | 16 [7 to 100]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the duration of time from start of treatment to time of recurrence, progression, or death due to any cause, whichever occurs first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LY3023414
Number analyzed (Participants) | 28
months | 2.5 [1.2 to 3.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: To determine the duration of response (DOR) of LY3023414 therapy, defined as the time from which measurement criteria are met for CR or PR (whichever status is recorded first) until the first date of documented disease progression.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | LY3023414
Number analyzed (Participants) | 28
months | 4.2 [1.4 to 9.6]

5. Secondary Outcome: Number of Participants Assessed for AE's With PI3K Activated Recurrent/Persistent Endometrial Cancer
Description: To assess the safety profile and tolerability of LY3023414 therapy in patients with PI3K activated recurrent/persistent endometrial cancer using the e current version of the National Cancer Institute Common Terminology Criteria for Adverse Events, which was version 4.03.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | LY3023414
Number analyzed (Participants) | 28
Participants | 28

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | LY3023414
All-Cause Mortality (participants affected / at risk) | 16/28
Serious Adverse Events (participants affected / at risk) | 7/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LY3023414 (N=28)
Alanine aminotransferase increased (Investigations) | 1
Allergic reaction (Immune system disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Cardiac troponin I increased (Investigations) | 1
Chills (General disorders) | 1
Creatinine increased (Investigations) | 1
Death NOS (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LY3023414 (N=28)
Alanine aminotransferase increased (Investigations) | 17
Alkaline phosphatase increased (Investigations) | 13
Anemia (Blood and lymphatic system disorders) | 25
Aspartate aminotransferase increased (Investigations) | 12
Constipation (Gastrointestinal disorders) | 8
Creatinine increased (Investigations) | 6
Fatigue (General disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 24
Hypoalbuminemia (Metabolism and nutrition disorders) | 20
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 14
Hyponatremia (Metabolism and nutrition disorders) | 12
Lymphocyte count decreased (Investigations) | 21
Nausea (Gastrointestinal disorders) | 13
Platelet count decreased (Investigations) | 16
White blood cell decreased (Investigations) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT02549989/Prot_SAP_000.pdf